CLINICAL TRIAL: NCT00979108
Title: The Value of Mechanical Traction in the Treatment of Cervical Radiculopathy
Brief Title: The Value of Traction in the Treatment of Cervical Radiculopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other); 59th Medical Wing (U.S. Federal Agency); Empi, A DJO Company (Industry)
Responsible Party: Principal Investigator, Shauna Bruun, Research Operations Coordinator, Intermountain Health Care, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1009133
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Radiculopathy; Neck Pain; Spinal Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Intervertebral Disk Displacement
Keywords: Radiculopathy; Neck pain; Physical therapy modalities; Rehabilitation
MeSH Terms: conditions — Radiculopathy; Neck Pain; Spinal Diseases; Musculoskeletal Diseases; Neuromuscular Diseases; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard exercise (Active Comparator): Subjects will be instructed in neck and postural exercises.
  Interventions: Other: Physical therapy rehabilitation
- Over-door traction and exercise. (Experimental): Subjects will receive traction utilizing an over-the-door traction unit in addition to neck and postural exercises.
  Interventions: Other: Physical therapy rehabilitation
- Mechanical traction and exercise (Experimental): Mechanical cervical traction will be utilized in addition to neck and postural exercises.
  Interventions: Other: Physical therapy rehabilitation

INTERVENTIONS:
Other: Physical therapy rehabilitation — Mechanical cervical traction will be applied at a moderate force and adjusted based on symptom relief. In addition, subjects will be trained in cervical and postural exercises.
  Other Names: Saunders 3D Active Trac
  Arms: Mechanical traction and exercise
Other: Physical therapy rehabilitation — Subjects will be instructed in use of an over-the-door traction unit utilizing weights up to 20 pounds in sitting. In addition, subjects will be trained in neck and postural exercises.
  Arms: Over-door traction and exercise.
Other: Physical therapy rehabilitation — Subjects will be instructed in neck and postural exercises.
  Arms: Standard exercise

SUMMARY:
The purpose of this study is to determine the effectiveness of adding mechanical traction to standard physical therapy treatments for patients with neck and arm pain.

DETAILED DESCRIPTION:
Cervical traction is an intervention frequently recommended for the treatment of patients with neck pain. Systematic reviews have not endorsed the use of mechanical traction for patients with neck pain, however these reviews note the poor methodological quality of available research. Trials that have been performed have examined heterogeneous samples of patients with neck pain. It may be that cervical traction has not shown to be effective because only a specific subgroup may benefit from it. Most experts believe that traction is most beneficial for individuals with neck pain extending into the upper extremity who have signs of nerve root compression. Randomized clinical trials examining the effectiveness of traction for patients with these specific characteristics have not been performed. Preliminary studies support the hypothesis that there exists a specific subgroup of patients with neck pain likely to benefit from traction

The current study will address 3 important questions:

1. Will the existence of a more specific subgroup of patients who benefit from traction along with a standard exercise program be validated in a second sample of patients?
2. Is cervical traction a critical component of the treatment necessary to maximize outcomes for patients in this subgroup?
3. Do two commonly used traction protocols differ in their effectiveness for patients in this subgroup? (Specifically, we study will compare supine mechanical traction to over-the-door traction.)

ELIGIBILITY:
Inclusion Criteria:

1. Primary complaint of neck pain with symptoms (pain and/or numbness) extending distal to the acromioclavicular joint or caudal to the superior border of the scapula (may be unilateral or bilateral).
2. Age between 18-70 years old
3. Neck Disability Score score >10 points

Exclusion Criteria:

1. Red flags indicative of a serious or non-musculoskeletal condition (i.e. tumor, fracture, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, etc.)
2. Diagnosis of cervical spinal stenosis based on CT or MRI imaging
3. Evidence of cervical myelopathy or central nervous system involvement, (e.g., hyperreflexia, intrinsic muscle wasting of the hands, unsteadiness during gait, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, presence of pathologic reflexes (i.e. positive Hoffman's or Babinski reflex).
4. Prior surgery to the neck or thoracic spine
5. Inability to comply with treatment and follow-up schedule

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Neck Disability Questionnaire | Baseline, 4 weeks, 6 months, 1year

SECONDARY OUTCOMES:
Global Rating of Change | Baseline, 4 weeks, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fritz, Principal Investigator — IHC Health Services, Inc., Dba: TOSH
Locations (2):
- United States (2):
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Intermountain Healthcare, Rehab Agency, Salt Lake City, Utah

REFERENCES:
- [Result] Fritz JM, Thackeray A, Brennan GP, Childs JD. Exercise only, exercise with mechanical traction, or exercise with over-door traction for patients with cervical radiculopathy, with or without consideration of status on a previously described subgrouping rule: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Feb;44(2):45-57. doi: 10.2519/jospt.2014.5065. Epub 2014 Jan 9. PMID 24405257